CLINICAL TRIAL: NCT04186754
Title: Interdisciplinary Randomized Study of an Integral Respiratory Rehabilitation Program in Oncological Patient With Disney
Brief Title: Study of an Integral Respiratory Rehabilitation Program in Oncological Patient With Disney
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 245380
Record Dates: First submitted 2019-09-03; First posted 2019-12-05 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Occupational Therapy; Cancer; Dyspnea; Rehabilitation
Keywords: Occupational Therapy; Cancer; Dyspnea
MeSH Terms: conditions — Neoplasms; Dyspnea | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive functional care plan (Experimental): The intervention will be carried out thanks to the "reeducation to the effort" carried out in the individuals, which will have the following interventions:
  The treatment should be carried out INDIVIDUALIZED, in the hospital room or in a conditioned room, in sessions of approximately 30 minutes and on a daily basis. Carried out by professionals in the disciplines of nursing and occupational therapy.
  Interventions: Procedure: Comprehensive functional care plan
- Traditional intervention without rehabilitation (Active Comparator): * Nursing care.
  * Medical care.
  * Spiritual attention.
  Interventions: Procedure: Traditional intervention without rehabilitation

INTERVENTIONS:
Procedure: Comprehensive functional care plan — The treatment should be carried out INDIVIDUALIZED, in the hospital room or in a conditioned room, in sessions of approximately 30 minutes and on a daily basis. Carried out by professionals in the disciplines of nursing and occupational therapy.
  Arms: Comprehensive functional care plan
Procedure: Traditional intervention without rehabilitation — Clinical control by nursing professionals and exclusively pharmacological treatment
  Arms: Traditional intervention without rehabilitation

SUMMARY:
Hypothesis: Oncological patients presenting with respiratory problems will benefit both at a functional level and at a level of quality of life from the inclusion of a program of integral respiratory rehabilitation from the perspective of nursing and occupational therapy at the time of admission hospital for an exacerbation of his respiratory symptoms.

Main objective: to verify the effectiveness of a comprehensive respiratory rehabilitation program carried out from the perspective of an interdisciplinary team made up of nurses, occupational therapists and doctors in the improvement of the respiratory problem referred to oncological disease.

Design: experimental, randomized, stratified, longitudinal prospective study through a parallel scheme of fixed assignment with experimental group and control group.

DETAILED DESCRIPTION:
Hypothesis: Oncological patients presenting with respiratory problems will benefit both at a functional level and at a level of quality of life from the inclusion of a program of integral respiratory rehabilitation from the perspective of nursing and occupational therapy at the time of admission hospital for an exacerbation of his respiratory symptoms.

Main objective: to verify the effectiveness of a comprehensive respiratory rehabilitation program carried out from the perspective of an interdisciplinary team made up of nurses, occupational therapists and doctors in the improvement of the respiratory problem referred to oncological disease.

Design: experimental, randomized, stratified, longitudinal prospective study through a parallel scheme of fixed assignment with experimental group and control group.

Location: Medical Oncology Service of the University Hospital of Salamanca.

PROCESS

The study will be carried out in accordance with the provisions of the Medical Oncology Service of the University Hospital of Salamanca.

Prior authorization by the patient after informed consent read, understood and signed will proceed to randomization. The subjects will be assigned prospectively, to the study, through a randomization process, using random numbers generated by computer, to the two conditions of the study: Control condition: Group I and Experimental condition: Group II.

In the generated table, those individuals that correlate with an odd number will be assigned to the control condition, while on the contrary, those with even numbers will correspond to the experimental group.

In the first, the control group will proceed to carry out an exhaustive evaluation at the time of admission and at the time of discharge, which will consist of: BODE index, which measures muscle mass index (BMI), dyspnea level by Medical Research Council scale, exercise capacity by 6-minute walk test and forced expiratory volume during the first second (FEV1); With all this data the investigators will establish a score in this index. The investigators will also value activities of daily living (AVD), thanks to the BARTHEL index and Health Related Quality of Life (HRQOL) thanks to the EuroQol-5D.

Finally, the investigators will take into account a series of intervening variables collected in a database, previously prepared solely and exclusively for the realization of this project.

In the second, the experimental group, in addition to performing the same assessment, upon admission and discharge, as in the control group, will be carried out with each individual sessions of Integral Respiratory Rehabilitation, by professionals from the disciplines of nursing and occupational therapy, on a daily basis with an approximate duration of 30-45 minutes.

INTEGRAL RESPIRATORY REHABILITATION PROGRAM

The work methodology used will follow the theoretical basis of Rehabilitation based on functional integration. It is a new method of intervention in patients in acute and subacute phase, based fundamentally on "treating dysfunction with function".

It emerged to respond to the continuing demands of patients and caregivers in the geriatric service, oriented towards the need to achieve greater patient independence. There was a demotivation of the patients towards the performance of conventional therapeutic treatments focused on the deficit. For this, it was necessary to create a new intervention method that would achieve the greatest possible functionality in the shortest period of time (stays in very mild acute units), seeking much more effective, fast and dynamic treatments.

Functional mobility will be the central axis of the treatment. With this type of intervention, the reinforcement of the patient's functional gain will be immediate, so that both he and his family / caregiver will be more involved with the treatment. It can be said that the level of collaboration increases, ensuring that during the rest of the day, in which the patient does not receive interventions, the benefits obtained continue to be enhanced (this is what the investigators call 24-hour therapy), stimulating and mobilizing the patient outside of the room (wandering around, in a wheelchair ...) taking it to the bathroom, letting them eat alone ... in short, promoting their independence and preventing the respiratory patient cycle from being fulfilled, which will lead to loss of functionality resulting from dyspnea that will secondarily worsen the quality of individual's life

The intervention will be carried out thanks to the "reeducation to the effort" carried out in the individuals, which will have the following interventions:

* Progressive mobilization.
* Gradation and simplification of activities.
* Teaching energy saving techniques.
* Modification of daily activities.
* Breathing exercises.
* Airway permeabilization techniques.

ELIGIBILITY:
Inclusion Criteria:

* Have an anatomopathological diagnosis of cancer disease among the reasons for admission.
* Present at least some level 2 or moderate dyspnea parameters on the MRC scale.
* Be admitted to the University Hospital of Salamanca.
* Sign an informed consent authorizing their voluntary participation in the study.

Exclusion Criteria:

* Present a diagnosis of bone metastases.
* Not having an adequate cognitive state to understand and carry out the orders provided.
* Carry out a number of rehabilitation sessions of less than 5.
* Present hemoglobin levels below 10g / dl.
* To be an active smoker today.
* Present pleural effusion.
* Present febrile neutropenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Dyspnoea | Up to 3 years
  MRC scale

SECONDARY OUTCOMES:
Activities of Daily Living | Up to 3 years
  Barthel index

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo IP Fernández, OT, Principal Investigator — University of Salamanca
Locations (1):
- Eduardo José Fernández, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
A specific database will be created to which any external researcher can access after contact by email to the email edujfr@usal.es
Time Frame: We do not establish a specific period of time, access will be permanent.
Access Criteria: Researcher upon invitation by mail

REFERENCES:
- [Derived] Fernandez-Rodriguez EJ, Sanchez-Gomez C, Fonseca-Sanchez E, Cruz-Hernandez JJ, Rihuete-Galve MI. Impact of a multimodal effort re-education programme on functionality, physical performance, and functional capacity in cancer patients with dyspnoea: a randomised experimental study. Support Care Cancer. 2024 Sep 6;32(10):639. doi: 10.1007/s00520-024-08852-1. PMID 39237780